CLINICAL TRIAL: NCT01499888
Title: Phase I/II Study of Allogeneic Stem Cell Transplantation to Treat Clinically Aggressive Sickle Cell Disease (SCD)
Brief Title: Ph I/II Study of Allogeneic SCT for Clinically Aggressive Sickle Cell Disease (SCD)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0096
Record Dates: First submitted 2011-11-23; First posted 2011-12-26 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Subtype Hgb SS; Subtype Hgb SC; Subtype Hgb SB; Chronic Transfusion Therapy; Prior Stroke; Allogeneic; Stem Cell Transplantation; Alemtuzumab; Sirolimus; Total Body Irradiation; Hydroxyurea Intolerant
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic Non-Myeloablative Stem Cell Transplantation (Experimental): The transplant regimen will consist of alemtuzumab 1mg/kg divided over five days, 300 cGy TBI, followed by sirolimus dosed for a target serum trough level of 10- 15 ng/mL.
  Interventions: Procedure: Allogeneic Non-Myeloablative Stem Cell Transplantation; Drug: Alemtuzumab; Drug: Sirolimus

INTERVENTIONS:
Procedure: Allogeneic Non-Myeloablative Stem Cell Transplantation — Alemtuzumab-based non-myeloablative allogeneic hematopoietic stem cell transplantation using immune-suppressive agents and low-dose total body irradiation (TBI) without standard chemotherapy.
  Transplant regimen Day -7 to -3: Alemtuzumab (1mg/kg, total dose) divided over the 5 days, IVPB over 2 hours daily Day -3 until 100% chimerism obtained: Sirolimus dosed for target trough level of 10-15 ng/mL Day -2: Total body irradiation with 300cGy Day 0: Stem cell infusion
Drug: Alemtuzumab — In this protocol, patients will be given alemtuzumab 1mg/kg divided equally over five days with the maximum dose of 20mg per day.
  Other Names: Campath; MabCampath; Campath-1H
Drug: Sirolimus — On day -1, patients will receive a loading dose of 12 mg followed by 4 mg per day. Subsequent dosing will be based on clinical toxicity, GVHD concurrent medications, medical conditions, prior drug levels, drug-drug interactions, and blood levels with target of 3 to 12 ng/mL.
  Other Names: Rapamune; Rapamycin

SUMMARY:
The investigators propose to determine the engraftment and transplant related morbidity and mortality after a non-myeloablative allogeneic hematopoietic stem cell transplant protocol using immune- suppressive agents and low-dose total body irradiation (TBI) without standard chemotherapy in patients with aggressive sickle cell disease who are not candidates for or experienced complications from hydroxyurea therapy.

Fully HLA matched siblings will be used as donors for hematopoietic stem cells to reduce the risk of morbidity and mortality in this cohort of patients.

DETAILED DESCRIPTION:
Sickle cell disease is an inherited defect caused by a mutation in the Beta globin gene affecting red blood cells. Symptoms begin at 6 months of life and often lead to debilitating vaso-occlusive pain crises, acute insults to vital organ systems,chronic organ injury, and decreased survival with median survival estimated at 42 years for men and 48 years for women. Several cohort studies have identified clinical and laboratory predictors for decreased survival which include acute complications, and chronic complications of sickle cell disease.

Hydroxyurea is the only FDA approved drug to help ameliorate symptoms associated with sickle cell disease. Two nonrandomized studies have suggested a reduction in mortality after 17 years of long term hydroxyurea treatment. However, the mortality rate is still high in the hydroxyurea cohort at 43.1% and only 38.1% of patients have a rise in fetal hemoglobin indicating that a significant percentage of patients still have aggressive disease despite hydroxyurea treatment. Hydroxyurea therapy also does not seem to prevent the development of pulmonary hypertension.

In the pediatric population, patients that have not clinically improved despite optimized hydroxyurea management are offered allogeneic stem cell transplantation. Until recently, the options were more limited in adults with sickle cell disease that had aggressive disease despite hydroxyurea therapy. Most rely on chronic red blood cell transfusions which carry significant risks of infection, iron overload, and alloimmunization. Up to 50% of patients with sickle cell disease who are on chronic transfusion therapy will develop allo-antibodies making further transfusions difficult with a high potential for hemolytic transfusion reactions.

Patients with sickle cell disease often have chronic underlying organ disease and so the effects of chemotherapy may be unpredictable and potentially more harmful, making low dose TBI more attractive as a safer modality for conditioning.

The investigators propose to determine the engraftment and transplant related morbidity and mortality after a non-myeloablative allogeneic hematopoietic stem cell transplant protocol using immune- suppressive agents and low-dose total body irradiation (TBI) without standard chemotherapy in patients with aggressive sickle cell disease who are not candidates for or experienced complications from hydroxyurea therapy.

Fully HLA matched siblings will be used as donors for hematopoietic stem cells to reduce the risk of morbidity and mortality in this cohort of patients.

An optional correlative trial will be conducted to compare ocular findings after stem cell transplantation with those findings before stem cell transplantation. Anterior and posterior ocular examination as well as objective tests will be performed on subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease, subtype Hgb SS, SC, or SB disease who are on chronic transfusion therapy for a prior stroke or those patients who were intolerant of hydroxyurea therapy or were being treated with hydroxyurea therapy and were complicated by at least one of the following:

  * Stroke or central nervous system event lasting longer than 24 hours
  * Frequent vaso-occlusive pain episodes, defined as ≥ 3 per year severe enough to interfere with the patient's normal daily function or require medical attention in the clinic, emergency room, acute care center, or hospital
  * Recurrent episodes of priapism, defined as ≥ 2 per year requiring emergency room visits
  * Acute chest syndrome with recurrent hospitalizations, defined as ≥ 2 lifetime events
  * Red-cell alloimmunization (≥ 2 antibodies) during longterm transfusion therapy
  * Bilateral proliferative retinopathy with major visual impairment in at least one eye
  * Osteonecrosis of 2 or more joints
  * Sickle cell nephropathy
  * Stage I or II sickle lung disease
  * Symptoms of pulmonary hypertension and mean pulmonary artery pressure > 25mmHg
* Age 16-60 years
* Karnofsky performance status of 70 or higher
* Adequate cardiac function, defined as left ventricular ejection fraction ≥ 40%
* Adequate pulmonary function, defined as diffusion lung capacity of carbon monoxide ≥ 50%
* Estimated GFR ≥ 30mL/min as calculated by the modified MDRD equation
* ALT ≤ 3x upper limit of normal
* No evidence of chronic active hepatitis or cirrhosis
* HIV-negative
* Patient is not pregnant
* History of compliance with medications and medical care
* Patient is able and willing to sign informed consent
* Patient has an HLA-identical matched related donor

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2028-09-23 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
To determine the engraftment after non-myeloablative HSC transplant | Up to 30 days post-transplant.

SECONDARY OUTCOMES:
To assess the frequency of acute and chronic complications of sickle cell disease | Up to 100 days post-transplant.
  To assess for the frequency of acute and chronic complications of sickle cell disease after allogeneic hematopoietic stem cell transplantation using a protocol of immunosuppressive agents and low-dose TBI without standard chemotherapy. The acute complications include vaso-occlusive pain episodes, acute chest syndrome, stroke, and priapism. The chronic complications include nephropathy, retinopathy, osteonecrosis, pulmonary artery pressures, and chronic lung disease.
To evaluate the immune reconstitution after transplant. | Up to 12 months after transplant.
To determine the transplant related morbidity and mortality. | Up to 365 days post-transplant.
  Transplant related mortality will be evaluated at day 100 and day 365. If mortality is greater than 25% at day 100 or 35% at day 365, then the trial will be closed.
To determine the long-term engraftment after non-myeloablative HSC transplant | Up to 10 years post-transplant.

OTHER OUTCOMES:
To determine whether ocular findings from sickle cell disease are reversible in patients undergoing stem cell transplantation to treat their sickle cell disease. | Up to 5 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States